CLINICAL TRIAL: NCT03070873
Title: Anatomical and Functional Outcomes of Perigee and Apogee Mesh in Total Pelvic Floor Reconstruction Versus Gynecare Prolift
Acronym: mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xirong Guo, Vice president of Obstetrics and Gynecology Hospital Affiliated to Nanjing Medical University, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: NMU-201666
Record Dates: First submitted 2017-02-15; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: Quality of life; Vaginal mesh; Mesh complications
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: The investigators divided the patients randomly into three groups:
  The group A was a total of 91 patients who accepted transvaginal hysterectomy and total pelvic floor reconstruction combined Perigee and Apogee polypropylene mesh(PA)；
  The group B was a total of 97 patients who accepted transvaginal hysterectomy and total pelvic floor reconstruction with Gynecare prolift polypropylene mesh；
  The group C was a total of 70 patients who accepted transvaginal hysterectomy and anterior and posterior vaginal wall repair without any mesh.
Who Masked: Participant, Investigator
Masking Description: In the study the operation was performed by three surgeons, the patients received surgery by the doctor when the patients saw in the outpatient clinic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- group A (Experimental): accepted Perigee and Apogee mesh(PA)
  Interventions: Device: Perigee and Apogee Mesh
- group B (Experimental): accepted Gynecare prolift mesh
  Interventions: Device: Gynecare Prolift Mesh
- group C (Placebo Comparator): Traditional surgery without any mesh
  Interventions: Procedure: Traditional Surgery

INTERVENTIONS:
Device: Perigee and Apogee Mesh — The investigators divided the patients randomly into three groups :the group A received Perigee and Apogee polypropylene mesh(PA)；the group B received Gynecare prolift polypropylene mesh；the group C was without any mesh.
  Arms: group A
Device: Gynecare Prolift Mesh — The investigators divided the patients randomly into three groups :the group A received Perigee and Apogee polypropylene mesh(PA)；the group B received Gynecare prolift polypropylene mesh；the group C was without any mesh.
  Arms: group B
Procedure: Traditional Surgery — The investigators divided the patients randomly into three groups :the group A received Perigee and Apogee polypropylene mesh(PA)；the group B received Gynecare prolift polypropylene mesh；the group C was without any mesh.
  Arms: group C

SUMMARY:
The investigators designed a prospective study in this article to evaluate the efficacy, the life quality and the complications of two different meshes of type I (one is Perigee/Apogee, the other is named Gynecare prolift) versus traditional surgery, and also studied the influence of some surgical procedures on the prognosis.

DETAILED DESCRIPTION:
Pelvic organ prolapse is defined as a downward descent of the pelvic organs that results in the protrusion of vagina, uterus, or both. The investigators designed a prospective study in this article to evaluate the efficacy, the life quality and the complications of two different meshes of type I (one is Perigee/Apogee, the other is named Gynecare prolift) versus traditional surgery. The investigators also studied the influence of some surgical procedures on the prognosis. In this study，The investigators divided the patients randomly into three groups :the group A was a total of 91 patients who accepted transvaginal hysterectomy and total pelvic floor reconstruction combined Perigee and Apogee polypropylene mesh(PA)；the group B was a total of 97 patients who accepted transvaginal hysterectomy and total pelvic floor reconstruction with Gynecare prolift polypropylene mesh；the group C was a total of 70 patients who accepted transvaginal hysterectomy and anterior and posterior vaginal wall repair without any mesh.The investigators did POP-Q measurements and questionnaire preoperatively and postoperatively and recorded volume of bleeding，day of postoperative indwelling catheter and the mesh complications。

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage III ~ IV degree of anterior and posterior vaginal wall prolapse and uterine prolapse (total pelvic floor prolapse) by the Pelvic Organ Prolapse Quantification System (POP-Q) were included

Exclusion Criteria:

* Simple anterior or posterior wall prolapse, simple uterine prolapse, combined with stress urinary incontinence, overactive bladder (OAB), pelvic floor repair surgery history and recurrent patients
* Local or systemic conditions that would preclude surgery or affect healing such as restricted leg motion (inability to conform to the lithotomy position)
* Vaginal bleeding;coagulation disorders
* Infection,or uncontrolled hypertension and diabetes mellitus
* Pelvic cancer and radiation to the pelvic area in the previous 6 months.
* Also women of reproductive age, and planning of pregnancy were also excluded for mesh usage.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-01-30 (Actual); Study Completion 2014-01-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification | at 12 months after surgery
  the prolapse of stage II and above is defined as recurrence in POP-Q stage.
sexual quality of life through the pelvic organ prolapse / urinary incontinence sexual questionnaire | at 12 months after surgery
  PISQ-12
pelvic floor distress inventory short form | at 12 months after surgery
  PFDI-20
mesh exposure | at 12 months after surgery
  mesh was seen in the vagina by gynecological examination
sexual quality of life through the pelvic organ prolapse / urinary incontinence sexual questionnaire | at 24 months after surgery
  PISQ-12
Pelvic Organ Prolapse Quantification | at 24 months after surgery
  the prolapse of stage II and above is defined as recurrence in POP-Q stage.
pelvic floor distress inventory short form | at 24 months after surgery
  PFDI-20
mesh exposure | at 24 months after surgery
  mesh was seen in the vagina by gynecological examination
sexual quality of life through the pelvic organ prolapse / urinary incontinence sexual questionnaire | baseline
  PISQ-12
pelvic floor distress inventory short form | baseline
  PFDI-20

SECONDARY OUTCOMES:
stress urinary incontinence | at 1 months after surgery
  leakage of urine with exertion or with sneezing or coughing
stress urinary incontinence | 3 months after surgery
  leakage of urine with exertion or with sneezing or coughing
Volume of bleeding | during the operation
Elevated blood pressure | during the operation
Day of postoperative indwelling catheter | 1 months after surgery
Number of constipation | 1 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Fei Shen, Study Director — director of Gynecology Department , Obstetrics and Gynecology Hospital Affiliated to Nanjing Medical University

IPD SHARING:
Plan to Share IPD: Yes